CLINICAL TRIAL: NCT00372229
Title: A Randomized Trial Comparing Valcyte CMV Prophylaxis Versus Pre-emptive Therapy After Renal Transplantation Using Proteomics for Monitoring of Graft Alteration
Brief Title: A Study of Valcyte (Valganciclovir) CMV Prophylaxis After Renal Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ML19313
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir; Ganciclovir

ARMS (2):
- Valganciclovir Cytomegalovirus (CMV) Prophylaxis (Experimental)
  Interventions: Drug: Valganciclovir CMV Prophylaxis
- Pre-emptive CMV Therapy (Active Comparator)
  Interventions: Drug: Valganciclovir (Pre-emptive CMV Therapy); Drug: Ganciclovir

INTERVENTIONS:
Drug: Valganciclovir CMV Prophylaxis — 900 mg valganciclovir, taken orally once daily, adjusted to renal function starting within 14 days of transplantation until Day 100 after transplantation.
  Other Names: Valcyte
  Arms: Valganciclovir Cytomegalovirus (CMV) Prophylaxis
Drug: Valganciclovir (Pre-emptive CMV Therapy) — If plasma polymerase chain reaction (PCR) ≥ 400 CMV copies/millilitre, then 1800 mg valganciclovir per day adjusted to renal function for at least 14 days until the second negative PCR (below 400 copies/ml) followed by secondary prophylaxis for 28 days with 900 mg valganciclovir adjusted to renal function. If CMV disease or no response to valganciclovir treatment after 14 days (not falling viral load), then intravenous (IV) ganciclovir or additional appropriate therapy could have been administered according to the local site's standard, instead of valganciclovir.
  Other Names: Valcyte
  Arms: Pre-emptive CMV Therapy
Drug: Ganciclovir — If CMV disease or no response to valganciclovir treatment after 14 days (not falling viral load), then intravenous (IV) ganciclovir or additional appropriate therapy could have been administered according to the local site's standard, instead of valganciclovir.
  Arms: Pre-emptive CMV Therapy

SUMMARY:
This 2 arm study will compare the efficacy of 100 days of Valcyte (900mg po daily) prophylaxis with that of no prophylaxis, under the condition of pre-emptive therapy of active CMV infection, in CMV positive renal transplant recipients. The influence of the two prevention concepts on the occurrence of direct and indirect effects of active CMV infections will be compared. The anticipated time on study treatment is 3 months-1 year, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary renal allograft within preceding 14 days;
* IgG seropositive for CMV;
* receiving immunosuppressive therapy.

Exclusion Criteria:

* active CMV infection;
* current/history of malignancy;
* acute steroid resistant rejection episode since transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2006-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Austria (2):
  - Innsbruck
  - Vienna
- Germany (20):
  - Aachen
  - Berlin
  - Bremen
  - Cologne
  - Düsseldorf
  - Erlangen
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
  - Hannoversch Münden
  - Hanover
  - Jena
  - Leipzig
  - Lübeck
  - München
  - Münster
  - Regensburg
  - Tübingen
  - Würzburg

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Mazzola P, Schaeffeler E, Witzke O, Nitschke M, Kliem V, Zortel M, Wagner EM, Schwab M, Hauser IA. No association of genetic variants in TLR4, TNF-alpha, IL10, IFN-gamma, and IL37 in cytomegalovirus-positive renal allograft recipients with active CMV infection-Subanalysis of the prospective randomised VIPP study. PLoS One. 2021 Apr 16;16(4):e0246118. doi: 10.1371/journal.pone.0246118. eCollection 2021. PMID 33861738
- [Derived] Witzke O, Nitschke M, Bartels M, Wolters H, Wolf G, Reinke P, Hauser IA, Alshuth U, Kliem V. Valganciclovir Prophylaxis Versus Preemptive Therapy in Cytomegalovirus-Positive Renal Allograft Recipients: Long-term Results After 7 Years of a Randomized Clinical Trial. Transplantation. 2018 May;102(5):876-882. doi: 10.1097/TP.0000000000002024. PMID 29166336

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 342 participants were screened, and 43 participants were not randomized. Central randomization stratified by study center and by induction immunosuppression with polyclonal antibodies, such as such as antithymocyte globuline (ATG), anti-lymphocyte globulin (ALG), or Muromonab-CD3 was performed.
Groups:
- Valganciclovir Cytomegalovirus (CMV) Prophylaxis: Valganciclovir (prophylaxis): 900 mg valganciclovir, taken orally once daily, adjusted to renal function starting within 14 days of transplantation until Day 100 after transplantation.
- Pre-emptive CMV Therapy: Valganciclovir (Pre-emptive CMV Therapy): If plasma polymerase chain reaction (PCR) ≥ 400 CMV copies/millilitre, then 1800 mg valganciclovir per day adjusted to renal function for at least 14 days until the second negative PCR (below 400 copies/ml) followed by secondary prophylaxis for 28 days with 900 mg valganciclovir adjusted to renal function.
  Ganciclovir: If CMV disease or no response to valganciclovir treatment after 14 days (not falling viral load), then intravenous (IV) ganciclovir or additional appropriate therapy could have been administered according to the local site's standard, instead of valganciclovir.
Period: Study Phase
Arm/Group | Valganciclovir Cytomegalovirus (CMV) Prophylaxis | Pre-emptive CMV Therapy
Started | 148 | 151
Completed | 117 | 122
Not Completed | 31 | 29
Not completed — Graft loss | 0 | 3
Not completed — Protocol Violation | 3 | 4
Not completed — Consent withdrawn | 16 | 14
Not completed — Refused treatment/did not cooperate | 3 | 1
Not completed — Death | 3 | 2
Not completed — Reason not specified | 3 | 2
Not completed — Lost to Follow-up | 3 | 3
Period: Follow-Up Phase
Arm/Group | Valganciclovir Cytomegalovirus (CMV) Prophylaxis | Pre-emptive CMV Therapy
Started | 117 | 122
Completed | 71 | 70
Not Completed | 46 | 52
Not completed — Graft loss | 8 | 7
Not completed — Consent withdrawn | 13 | 19
Not completed — Refused treatment/did not cooperate | 0 | 1
Not completed — Adverse event/intercurrent illness | 1 | 0
Not completed — Death | 9 | 12
Not completed — Administrative | 1 | 0
Not completed — Reason not specified | 2 | 3
Not completed — Lost to Follow-up | 12 | 10

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized participants.
Groups:
- Valganciclovir CMV Prophylaxis: Valganciclovir (prophylaxis): 900 mg valganciclovir, taken orally once daily, adjusted to renal function starting within 14 days of transplantation until Day 100 after transplantation.
- Total: Total of all reporting groups
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy | Total
Number analyzed (Participants) | 148 | 151 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.18 (13.463) | 54.24 (11.906) | 52.73 (12.771)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 55 | 100
  Male | 103 | 96 | 199

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Active Cytomegalovirus (CMV) Infection Within 12 Months
Description: Active CMV infection was defined as plasma polymerase chain reaction (PCR) ≥ 400 copies/millilitre (ml).
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number (96% Confidence Interval); unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 14.1 [7.0 to 21.1] | 42.6 [33.9 to 51.3]
Statistical Analysis 1: Comparison: Valganciclovir CMV Prophylaxis vs Pre-emptive CMV Therapy; Test type: Superiority or Other; Difference = -28.5, 96% CI 2-sided [-39.7 to -17.3], Standard Error of Mean 5.45

2. Primary Outcome: Percentage of Participants With CMV Disease Within 12 Months Including CMV Syndrome and Tissue Invasive Disease
Description: CMV disease comprises the two components of CMV syndrome as well as CMV tissue invasive disease. CMV syndrome was defined as viremia according to plasma PCR ≥ 400 copies/ml and at least one of the following signs: fever of ≥38 °C; new or increased malaise (malaise defined as normal activity reduced >50%; cannot work or unable to care for self; leukopenia on 2 successive measurements separated by at least 24 hours thrombocytopenia; elevation of hepatic transaminases (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) to at least 2 x upper limit of normal (ULN). CMV tissue invasive disease was defined as viremia according plasma PCR ≥ 400 copies/ml and clinical evidence of localized CMV infection (CMV inclusion cells or in situ detection of CMV antigen or deoxyribonucleic acid [DNA] by immunostaining or hybridization, respectively), cerebral spinal fluid [CSF]) and/or relevant symptoms or signs of organ dysfunction.
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number (96% Confidence Interval); unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 5.6 [1.4 to 9.8] | 16.9 [10.3 to 23.6]
Statistical Analysis 1: Comparison: Valganciclovir CMV Prophylaxis vs Pre-emptive CMV Therapy; Test type: Superiority or Other; Difference = -11.3, 96% CI 2-sided [-19.2 to -3.4], Standard Error of Mean 3.83

3. Primary Outcome: Urine Proteomic Pattern at Month 12
Description: Proteomics is the complete set of proteins expressed by an organism, tissue, or cell. Urine proteomic pattern was measured on a scale between -1, indicating no graft alteration, and +1, indicating graft alteration.
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
units on a scale | -0.1057 (0.1538) | 0.1452 (0.1006)
Statistical Analysis 1: Comparison: Valganciclovir CMV Prophylaxis vs Pre-emptive CMV Therapy; Test type: Superiority or Other; p = 0.1739, F-test; Mean Difference (Final Values) = 0.2509, 99% CI 2-sided [-0.2271 to 0.7289], Standard Error of Mean 0.1838

4. Primary Outcome: Percentage of Participants With Graft Loss at Month 84
Time Frame: Up to 84 months
Population: The intent-to-treat (ITT) population included all randomized participants. Descriptive analysis only.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 7.43 | 8.61

5. Secondary Outcome: Percentage of Participants With CMV Syndrome Within 12 Months
Description: CMV syndrome was defined as viremia according to plasma PCR ≥ 400 copies/ml and at least one of the following signs: fever of ≥38 °C; new or increased malaise (malaise defined as normal activity reduced >50%; cannot work or unable to care for self; leukopenia on 2 successive measurements separated by at least 24 hours thrombocytopenia; elevation of hepatic transaminases (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) to at least 2 x upper limit of normal (ULN).
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 5.6 [1.6 to 9.7] | 14.6 [8.7 to 20.6]

6. Secondary Outcome: Percentage of Participants With CMV Tissue Invasive Disease Within 12 Months
Description: CMV tissue invasive disease was defined as viremia: PCR ≥ 400 copies/ml and clinical evidence of localized CMV infection (CMV inclusion cells or in situ detection of CMV antigen or deoxyribonucleic acid [DNA] by immunostaining or hybridization, respectively), cerebral spinal fluid [CSF]) and/or relevant symptoms or signs of organ dysfunction.
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 3.3 [0.1 to 6.4] | 3.6 [0.5 to 6.8]

7. Secondary Outcome: Time to Occurrence of First Viremia Within 12 Months
Description: Viremia was defined as plasma PCR ≥ 400 copies/ml.
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
days | NA [NA to NA] — Median and confidence limits were not reached. | NA [160 to NA] — Median and upper confidence limit were not reached.

8. Secondary Outcome: Viral Burden at Viremia
Description: Time-weighted area under the curve (AUC) of the polymerase chain reaction (PCR). Viremia was defined as plasma PCR ≥ 400 copies/ml.
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Mean (Standard Deviation); unit: copies/ml*days
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
copies/ml*days | 5309.83 (14355.836) | 3765.8 (8480.521)

9. Secondary Outcome: Creatinine Clearance at Month 12
Description: Creatinine clearance was estimated using the Cockcroft-Gault formula.
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Mean (Standard Deviation); unit: millilitre(s)/minute
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
millilitre(s)/minute | 61.1 (23.30) | 61.3 (22.24)

10. Secondary Outcome: Percentage of Participants With at Least One Treated and Biopsy-Proven Acute Rejection Episode Within 12 Months
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 18.2 | 13.2

11. Secondary Outcome: Days of Hospitalization
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Median (Full Range); unit: days
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
days | 26.5 [0 to 258] | 32 [0 to 221]

12. Secondary Outcome: Relationship Between Proteomics Pattern and Graft Survival
Description: Proteomics is the complete set of proteins expressed by an organism, tissue, or cell. The proteomics of CKD273, CMV, and nephropathy was measured on a scale between -1, indicating no graft alteration, and +1, indicating graft alteration.
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants. Only participants with data were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
score on a scale
  CKD273:Visit 6: With Graft Loss (n=1, 4): number analyzed (Participants) | 1 | 4
  CKD273:Visit 6: With Graft Loss (n=1, 4) | 0.400 (NA) — Only one participant had data. | 0.800 (0.2944)
  CKD273:Visit 6: Without Graft Loss (n=112, 110): number analyzed (Participants) | 112 | 110
  CKD273:Visit 6: Without Graft Loss (n=112, 110) | 0.371 (0.3578) | 0.379 (0.3499)
  CKD273:Visit 13: With Graft Loss (n=0, 1): number analyzed (Participants) | 0 | 1
  CKD273:Visit 13: With Graft Loss (n=0, 1) |  | 0.500 (NA) — Only one participant had data.
  CKD273:Visit 13: Without Graft Loss (n=102, 109): number analyzed (Participants) | 102 | 109
  CKD273:Visit 13: Without Graft Loss (n=102, 109) | 0.258 (0.3719) | 0.293 (0.3648)
  CKD273:Visit 15: With Graft Loss (n=2, 0): number analyzed (Participants) | 2 | 0
  CKD273:Visit 15: With Graft Loss (n=2, 0) | 0.600 (0.5657) |
  CKD273:Visit 15: Without Graft Loss (n=104, 102): number analyzed (Participants) | 104 | 102
  CKD273:Visit 15: Without Graft Loss (n=104, 102) | 0.270 (0.3793) | 0.326 (0.3618)
  CMV:Visit 6: With Graft Loss (n=1, 4): number analyzed (Participants) | 1 | 4
  CMV:Visit 6: With Graft Loss (n=1, 4) | -0.500 (NA) — Only one participant had data. | -0.300 (0.7616)
  CMV:Visit 6: Without Graft Loss (n=112, 110): number analyzed (Participants) | 112 | 110
  CMV:Visit 6: Without Graft Loss (n=112, 110) | 0.000 (0.9535) | -0.007 (0.8984)
  CMV:Visit 13: With Graft Loss (n=0, 1): number analyzed (Participants) | 0 | 1
  CMV:Visit 13: With Graft Loss (n=0, 1) |  | -0.300 (NA) — Only one participant had data.
  CMV:Visit 13: Without Graft Loss (n=102, 109): number analyzed (Participants) | 102 | 109
  CMV:Visit 13: Without Graft Loss (n=102, 109) | 0.036 (0.7976) | -0.048 (0.7614)
  CMV:Visit 15: With Graft Loss (n=2, 0): number analyzed (Participants) | 2 | 0
  CMV:Visit 15: With Graft Loss (n=2, 0) | 0.100 (0.7071) |
  CMV:Visit 15: Without Graft Loss (n=104, 102): number analyzed (Participants) | 104 | 102
  CMV:Visit 15: Without Graft Loss (n=104, 102) | -0.076 (0.6922) | -0.068 (0.7081)
  Nephropathy:Visit 6: With Graft Loss (n=1, 4): number analyzed (Participants) | 1 | 4
  Nephropathy:Visit 6: With Graft Loss (n=1, 4) | -0.500 (NA) — Only one participant had data. | 1.100 (0.9933)
  Nephropathy:Visit 6:Without Graft Loss (n=112,110): number analyzed (Participants) | 112 | 110
  Nephropathy:Visit 6:Without Graft Loss (n=112,110) | 0.107 (1.1784) | 0.086 (1.0489)
  Nephropathy:Visit 13: With Graft Loss (n=0, 1): number analyzed (Participants) | 0 | 1
  Nephropathy:Visit 13: With Graft Loss (n=0, 1) |  | -0.800 (NA) — Only one participant had data.
  Nephropathy:Visit 13:Without Graft Loss(n=102,109): number analyzed (Participants) | 102 | 109
  Nephropathy:Visit 13:Without Graft Loss(n=102,109) | -0.050 (1.0624) | 0.008 (1.0848)
  Nephropathy:Visit 15: With Graft Loss (n=2, 0): number analyzed (Participants) | 2 | 0
  Nephropathy:Visit 15: With Graft Loss (n=2, 0) | 1.350 (2.8991) |
  Nephropathy:Visit15: Without Graft Loss(n=104,102): number analyzed (Participants) | 104 | 102
  Nephropathy:Visit15: Without Graft Loss(n=104,102) | -0.007 (0.8535) | 0.102 (1.1221)

13. Secondary Outcome: Relationship Between Proteomics Pattern and Participant Survival
Description: as for outcome 12
Time Frame: Up to 12 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
score on a scale
  CKD273:Visit 6: Did not Survive (n=2, 1): number analyzed (Participants) | 2 | 1
  CKD273:Visit 6: Did not Survive (n=2, 1) | 0.400 (0.1414) | 0.500 (NA) — Only one participant had data.
  CKD273:Visit 6: Survived (n=111, 113): number analyzed (Participants) | 111 | 113
  CKD273:Visit 6: Survived (n=111, 113) | 0.371 (0.3591) | 0.393 (0.3570)
  CKD273:Visit 13: Did not Survive (n=1, 1): number analyzed (Participants) | 1 | 1
  CKD273:Visit 13: Did not Survive (n=1, 1) | 0.700 (NA) — Only one participant had data. | 0.500 (NA) — Only one participant had data.
  CKD273:Visit 13: Survived (n=101, 109): number analyzed (Participants) | 101 | 109
  CKD273:Visit 13: Survived (n=101, 109) | 0.253 (0.3711) | 0.293 (0.3648)
  CKD273:Visit 15: Did not Survive (n=0, 0): number analyzed (Participants) | 0 | 0
  CKD273:Visit 15: Survived (n=106, 102): number analyzed (Participants) | 106 | 102
  CKD273:Visit 15: Survived (n=106, 102) | 0.276 (0.3824) | 0.326 (0.3618)
  CMV:Visit 6: Did not Survive (n=2, 1): number analyzed (Participants) | 2 | 1
  CMV:Visit 6: Did not Survive (n=2, 1) | 1.150 (1.3435) | -0.900 (NA) — Only one participant had data.
  CMV:Visit 6: Survived (n=111, 113): number analyzed (Participants) | 111 | 113
  CMV:Visit 6: Survived (n=111, 113) | -0.025 (0.9374) | -0.010 (0.8927)
  CMV:Visit 13: Did not Survive (n=1, 1): number analyzed (Participants) | 1 | 1
  CMV:Visit 13: Did not Survive (n=1, 1) | 0.400 (NA) — Only one participant had data. | -0.300 (NA) — Only one participant had data.
  CMV:Visit 13: Survived (n=101, 109): number analyzed (Participants) | 101 | 109
  CMV:Visit 13: Survived (n=101, 109) | 0.033 (0.8008) | -0.048 (0.7614)
  CMV:Visit 15: Did not Survive (n=0, 0): number analyzed (Participants) | 0 | 0
  CMV:Visit 15: Survived (n=106, 102): number analyzed (Participants) | 106 | 102
  CMV:Visit 15: Survived (n=106, 102) | -0.073 (0.6894) | -0.068 (0.7081)
  Nephropathy:Visit 6: Did not Survive (n=2, 1): number analyzed (Participants) | 2 | 1
  Nephropathy:Visit 6: Did not Survive (n=2, 1) | 0.150 (0.0707) | -0.100 (NA) — Only one participant had data.
  Nephropathy:Visit 6: Survived (n=111, 113): number analyzed (Participants) | 111 | 113
  Nephropathy:Visit 6: Survived (n=111, 113) | 0.101 (1.1851) | 0.124 (1.0640)
  Nephropathy:Visit 13: Did not Survive (n=1, 1): number analyzed (Participants) | 1 | 1
  Nephropathy:Visit 13: Did not Survive (n=1, 1) | 1.800 (NA) — Only one participant had data. | -0.800 (NA) — Only one participant had data.
  Nephropathy:Visit 13: Survived (n=101, 109): number analyzed (Participants) | 101 | 109
  Nephropathy:Visit 13: Survived (n=101, 109) | -0.068 (1.0514) | 0.008 (1.0848)
  Nephropathy:Visit 15: Did not Survive (n=0, 0): number analyzed (Participants) | 0 | 0
  Nephropathy:Visit 15: Survived (n=106, 102): number analyzed (Participants) | 106 | 102
  Nephropathy:Visit 15: Survived (n=106, 102) | 0.019 (0.9105) | 0.102 (1.1221)

14. Secondary Outcome: Proteomics Parameter: CKD273
Description: Proteomics is the complete set of proteins expressed by an organism, tissue, or cell. The proteomics of CKD273 was measured on a scale between -1, indicating no graft alteration, and +1, indicating graft alteration.
Time Frame: Up to 12 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
score on a scale
  Visit 6 (n=113, 114): number analyzed (Participants) | 113 | 114
  Visit 6 (n=113, 114) | 0.372 (0.3562) | 0.394 (0.3556)
  Visit 13 (n=102, 110): number analyzed (Participants) | 102 | 110
  Visit 13 (n=102, 110) | 0.258 (0.3719) | 0.295 (0.3637)
  Visit 15 (n=106, 102): number analyzed (Participants) | 106 | 102
  Visit 15 (n=106, 102) | 0.276 (0.3824) | 0.326 (0.3618)

15. Secondary Outcome: Proteomics Parameter: CMV
Description: Proteomics is the complete set of proteins expressed by an organism, tissue, or cell. The proteomics of CMV was measured on a scale between -1, indicating no graft alteration, and +1, indicating graft alteration.
Time Frame: Up to 12 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
score on a scale
  Visit 6 (n=113, 114): number analyzed (Participants) | 113 | 114
  Visit 6 (n=113, 114) | -0.004 (0.9504) | -0.018 (0.8927)
  Visit 13 (n=102, 110): number analyzed (Participants) | 102 | 110
  Visit 13 (n=102, 110) | 0.036 (0.7976) | -0.05 (0.7583)
  Visit 15 (n=106, 102): number analyzed (Participants) | 106 | 102
  Visit 15 (n=106, 102) | -0.073 (0.6894) | -0.068 (0.7081)

16. Secondary Outcome: Proteomics Parameter: Nephropathy
Description: Proteomics is the complete set of proteins expressed by an organism, tissue, or cell. The proteomics of nephropathy was measured on a scale between -1, indicating no graft alteration, and +1, indicating graft alteration.
Time Frame: Up to 12 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
score on a scale
  Visit 6 (n=113, 114): number analyzed (Participants) | 113 | 114
  Visit 6 (n=113, 114) | 0.102 (1.1745) | 0.122 (1.0595)
  Visit 13 (n=102, 110): number analyzed (Participants) | 102 | 110
  Visit 13 (n=102, 110) | -0.05 (1.0624) | 0.001 (1.0826)
  Visit 15 (n=106, 102): number analyzed (Participants) | 106 | 102
  Visit 15 (n=106, 102) | 0.019 (0.9105) | 0.102 (1.1221)

17. Secondary Outcome: Percentage of Participants Surviving at Month 12
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 98 | 98.7

18. Secondary Outcome: Percentage of Participants With Graft Survival at Month 12
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 98.6 | 96.0

19. Secondary Outcome: Percentage of Participants With Leukopenia Within 12 Months
Description: Leukopenia: white blood cell (WBC) of < 3,500/microlitre (μL) and < 1,000/μL
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 35.1 | 26.5

20. Secondary Outcome: Percentage of Participants With Neutropenia Within 12 Months
Description: Neutropenia: absolute neutrophil count (ANC) < 750/μL within 12 months.
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 16.9 | 12.6

21. Secondary Outcome: Percentage of Participants With Any Opportunistic Infection Within 12 Months
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants | 31.1 | 37.7

22. Secondary Outcome: Percentage of Participants With Post-Transplant Diabetes Mellitus
Time Frame: Up to 12 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants
  Month 6 | 2.7 | 1.3
  Month 12 | 3.4 | 0.7

23. Secondary Outcome: Percentage of Participants With Active CMV Infections Not Responding to Valganciclovir or IV Ganciclovir Treatment
Description: Active CMV infection was defined as plasma polymerase chain reaction (PCR) ≥ 400 copies/millilitre (ml).
Time Frame: Up to 12 months
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 17 | 82
percentage of participants | 11.8 | 18.3

24. Secondary Outcome: Number of Participants With CMV Viremia (Active CMV Infection) From Baseline to Month 24 and Every 12 Months up to Month 84
Description: Viremia (active CMV Infection) was defined as PCR ≥ 400 copies/ml.
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
Participants
  24 months | 16 | 59
  36 months | 16 | 59
  48 months | 16 | 59
  60 months | 16 | 59
  72 months | 17 | 60
  84 months | 17 | 60

25. Secondary Outcome: Number of Participants With CMV Disease From Baseline to Month 24 and Every 12 Months up to Month 84
Description: as for outcome 2
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
Participants
  24 months | 7 | 23
  36 months | 7 | 23
  48 months | 7 | 23
  60 months | 7 | 24
  72 months | 7 | 24
  84 months | 7 | 24

26. Secondary Outcome: Number of Participants With CMV Syndrome From Baseline to Month 24 and Every 12 Months up to Month 84
Description: as for outcome 5
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
Participants
  24 months | 7 | 20
  36 months | 7 | 20
  48 months | 7 | 20
  60 months | 7 | 21
  72 months | 7 | 21
  84 months | 7 | 21

27. Secondary Outcome: Number of Participants With CMV Tissue Invasive Disease From Baseline to Month 24 and Every 12 Months up to Month 84
Description: CMV tissue invasive disease was defined as viremia according plasma PCR ≥ 400 copies/ml and clinical evidence of localized CMV infection (CMV inclusion cells or in situ detection of CMV antigen or deoxyribonucleic acid [DNA] by immunostaining or hybridization, respectively), cerebral spinal fluid [CSF]) and/or relevant symptoms or signs of organ dysfunction.
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
Participants
  24 months | 4 | 5
  36 months | 4 | 5
  48 months | 4 | 5
  60 months | 4 | 5
  72 months | 4 | 5
  84 months | 4 | 5

28. Secondary Outcome: Number of Participants With Active CMV Infection After Month 24 and Every 12 Months up to Month 84
Description: Active CMV infection was defined as plasma polymerase chain reaction (PCR) ≥ 400 copies/millilitre (ml).
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
Participants
  24 months | 16 | 59
  36 months | 16 | 59
  48 months | 16 | 59
  60 months | 16 | 59
  72 months | 17 | 60
  84 months | 17 | 60

29. Secondary Outcome: Number of Participants With CMV Disease After Month 24 and Every 12 Months up to Month 84
Description: as for outcome 2
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
Participants
  24 months | 7 | 23
  36 months | 7 | 23
  48 months | 7 | 23
  60 months | 7 | 24
  72 months | 7 | 24
  84 months | 7 | 24

30. Secondary Outcome: Percentage of Participants Surviving at Month 24 and Every 12 Months up to Month 84
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants
  24 months | 97.97 | 94.70
  36 months | 95.95 | 94.04
  48 months | 94.59 | 93.38
  60 months | 92.57 | 92.05
  72 months | 90.54 | 89.40
  84 months | 90.54 | 88.74

31. Secondary Outcome: Number of Participants Who Died From Months 24 to Month 84
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
Participants
  24 months | 3 | 8
  36 months | 6 | 9
  48 months | 8 | 10
  60 months | 11 | 12
  72 months | 14 | 16
  84 months | 14 | 17

32. Secondary Outcome: Percentage of Participants With Graft Survival at Month 24 and Every 12 Months up to Month 84
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants
  24 months | 97.30 | 94.70
  36 months | 97.30 | 93.38
  48 months | 96.62 | 93.38
  60 months | 95.95 | 92.05
  72 months | 94.59 | 91.39
  84 months | 92.57 | 91.39

33. Secondary Outcome: Number of Participants Who Had Lost Their Transplant up to Month 84
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
Participants
  24 months | 4 | 8
  36 months | 4 | 10
  48 months | 5 | 10
  60 months | 6 | 12
  72 months | 8 | 13
  84 months | 11 | 13

34. Secondary Outcome: Number of Participants With Active CMV Infection Who Had Lost Their Transplant up to Month 84
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants. Only participants with active CMV infection were included in this analysis; 1 participant in each treatment arm had not developed active CMV infection until Month 72, and thus, they were only included in the number analyzed for results starting from that timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 17 | 60
Participants
  24 months: number analyzed (Participants) | 16 | 59
  24 months | 0 | 5
  36 months: number analyzed (Participants) | 16 | 59
  36 months | 0 | 7
  48 months: number analyzed (Participants) | 16 | 59
  48 months | 0 | 7
  60 months: number analyzed (Participants) | 16 | 59
  60 months | 0 | 9
  72 months | 0 | 9
  84 months | 1 | 9

35. Secondary Outcome: Number of Participants Without Active CMV Infection Who Had Lost Their Transplant up to Month 84
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants. Only participants without active CMV infection were included in this analysis; 1 participant in each treatment arm had not developed active CMV infection until Month 72, and thus, they were only included in the number analyzed for results before that timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 132 | 92
Participants
  24 months | 4 | 3
  36 months | 4 | 3
  48 months | 5 | 3
  60 months | 6 | 3
  72 months: number analyzed (Participants) | 131 | 91
  72 months | 8 | 4
  84 months: number analyzed (Participants) | 131 | 91
  84 months | 10 | 4

36. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants (With Versus Without Active CMV Infection) on Valganciclovir CMV Prophylaxis With First Occurrence of Graft Loss at Month 84
Description: An analysis for the time to first occurrence of graft loss within month 84 (by means of Kaplan-Meier analysis) was done for all patients who suffered at least once from acute CMV infection (CMV viremia) during this study versus all patients who did not suffer from acute CMV infection (CMV viremia) during the study. Active CMV infection was defined as plasma polymerase chain reaction (PCR) ≥ 400 copies/millilitre (ml).
Time Frame: Up to 84 months
Population: The intent-to-treat (ITT) population included all randomized participants. Only participants in the Valganciclovir CMV Prophylaxis arm (separated based on their active CMV infection status at Month 84) were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Valganciclovir CMV Prophylaxis,With CMV Infection at Month 84: Participants with active CMV infection at Month 84 that had received valganciclovir cytomegalovirus (CMV) prophylaxis. Valganciclovir (prophylaxis): 900 mg valganciclovir, taken orally once daily, adjusted to renal function starting within 14 days of transplantation until Day 100 after transplantation.
- Valganciclovir CMV Prophylaxis, No CMV Infection at Month 84: Participants without active CMV infection at Month 84 that had received valganciclovir cytomegalovirus (CMV) prophylaxis. Valganciclovir (prophylaxis): 900 mg valganciclovir, taken orally once daily, adjusted to renal function starting within 14 days of transplantation until Day 100 after transplantation.
Arm/Group | Valganciclovir CMV Prophylaxis,With CMV Infection at Month 84 | Valganciclovir CMV Prophylaxis, No CMV Infection at Month 84
Number analyzed (Participants) | 17 | 131
percentage of participants | 8.3 [0.0 to 24.0] | 11.5 [4.7 to 18.4]
Statistical Analysis 1: Comparison: Valganciclovir CMV Prophylaxis,With CMV Infection at Month 84 vs Valganciclovir CMV Prophylaxis, No CMV Infection at Month 84; Test type: Other — Descriptive analysis; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-20.2 to 13.9], Standard Error of Mean 8.71

37. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants (With Versus Without Active CMV Infection) on Pre-emptive CMV Therapy With First Occurrence of Graft Loss at Month 84
Description: as for outcome 36
Time Frame: Up to 84 months
Population: The intent-to-treat (ITT) population included all randomized participants. Only participants in the Pre-emptive CMV Therapy arm (separated based on their active CMV infection status at Month 84) were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pre-emptive CMV Therapy, With CMV Infection at Month 84; Pre-emptive CMV Therapy, No CMV Infection at Month 84: Participants with active CMV infection at Month 84 received valganciclovir pre-emptive CMV Therapy. Valganciclovir (Pre-emptive CMV Therapy): If plasma polymerase chain reaction (PCR) ≥ 400 CMV copies/millilitre, then 1800 mg valganciclovir per day adjusted to renal function for at least 14 days until the second negative PCR (below 400 copies/ml) followed by secondary prophylaxis for 28 days with 900 mg valganciclovir adjusted to renal function (If CMV disease or no response to valganciclovir treatment after 14 days (not falling viral load), then intravenous (IV) ganciclovir or additional appropriate therapy could have been administered according to the local site's standard, instead of valganciclovir).
Arm/Group | Pre-emptive CMV Therapy, With CMV Infection at Month 84 | Pre-emptive CMV Therapy, No CMV Infection at Month 84
Number analyzed (Participants) | 60 | 91
percentage of participants | 17.9 [7.2 to 28.6] | 5.8 [0.1 to 11.6]
Statistical Analysis 1: Comparison: Pre-emptive CMV Therapy, With CMV Infection at Month 84 vs Pre-emptive CMV Therapy, No CMV Infection at Month 84; Test type: Other — Descriptive analysis; Mean Difference (Final Values) = 12.1, 95% CI 2-sided [-0.1 to 24.2], Standard Error of Mean 6.21

38. Secondary Outcome: Number of Participants Who Had Lost Their Transplant or Died up to Month 84
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
Participants
  24 months | 7 | 15
  36 months | 9 | 18
  48 months | 12 | 19
  60 months | 16 | 23
  72 months | 21 | 28
  84 months | 24 | 29

39. Secondary Outcome: Percentage of Participants With Graft Survival or Participant Survival at Month 24 and Every 12 Months up to Month 84
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
percentage of participants
  24 months | 95.27 | 90.07
  36 months | 93.92 | 88.08
  48 months | 91.89 | 87.42
  60 months | 89.19 | 84.77
  72 months | 85.81 | 81.46
  84 months | 83.78 | 80.79

40. Secondary Outcome: Number of Participants With Graft Rejections by CMV Status (Positive or Negative) of the Donor at Month 24 and Every 12 Months up to Month 84
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
Participants
  24 months: CMV Positive Donor: number analyzed (Participants) | 91 | 79
  24 months: CMV Positive Donor: At Least One Rejection | 26 | 27
  24 months: CMV Positive Donor: No Rejections | 65 | 52
  24 months: CMV Negative Donor: number analyzed (Participants) | 57 | 72
  24 months: CMV Negative Donor: At Least One Rejection | 15 | 13
  24 months: CMV Negative Donor: No Rejections | 42 | 59
  36 months: CMV Positive Donor: number analyzed (Participants) | 91 | 79
  36 months: CMV Positive Donor: At Least One Rejection | 27 | 27
  36 months: CMV Positive Donor: No Rejections | 64 | 52
  36 months: CMV Negative Donor: number analyzed (Participants) | 57 | 72
  36 months: CMV Negative Donor: At Least One Rejection | 15 | 14
  36 months: CMV Negative Donor: No Rejections | 42 | 58
  48 months: CMV Positive Donor: number analyzed (Participants) | 91 | 79
  48 months: CMV Positive Donor: At Least One Rejection | 27 | 27
  48 months: CMV Positive Donor: No Rejections | 64 | 52
  48 months: CMV Negative Donor: number analyzed (Participants) | 57 | 72
  48 months: CMV Negative Donor: At Least One Rejection | 15 | 14
  48 months: CMV Negative Donor: No Rejections | 42 | 58
  60 months: CMV Positive Donor: number analyzed (Participants) | 91 | 79
  60 months: CMV Positive Donor: At Least One Rejection | 27 | 28
  60 months: CMV Positive Donor: No Rejections | 64 | 51
  60 months: CMV Negative Donor: number analyzed (Participants) | 57 | 72
  60 months: CMV Negative Donor: At Least One Rejection | 15 | 15
  60 months: CMV Negative Donor: No Rejections | 42 | 57
  72 months: CMV Positive Donor: number analyzed (Participants) | 91 | 79
  72 months: CMV Positive Donor: At Least One Rejection | 28 | 28
  72 months: CMV Positive Donor: No Rejections | 63 | 51
  72 months: CMV Negative Donor: number analyzed (Participants) | 57 | 72
  72 months: CMV Negative Donor: At Least One Rejection | 15 | 15
  72 months: CMV Negative Donor: No Rejections | 42 | 57
  84 months: CMV Positive Donor: number analyzed (Participants) | 91 | 79
  84 months: CMV Positive Donor: At Least One Rejection | 28 | 28
  84 months: CMV Positive Donor: No Rejections | 63 | 51
  84 months: CMV Negative Donor: number analyzed (Participants) | 57 | 72
  84 months: CMV Negative Donor: At Least One Rejection | 15 | 15
  84 months: CMV Negative Donor: No Rejections | 42 | 57

41. Secondary Outcome: Number of Graft Rejections by CMV Status (Positive or Negative) of the Donor at Month 24 and Every 12 Months up to Month 84
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants. The number analyzed in the table indicates the number of participants with at least one rejection episode at each timepoint.
Measure: Number; unit: graft rejections
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
graft rejections
  24 months: CMV Positive Donor: number analyzed (Participants) | 26 | 27
  24 months: CMV Positive Donor | 39 | 48
  24 months: CMV Negative Donor: number analyzed (Participants) | 15 | 13
  24 months: CMV Negative Donor | 20 | 27
  36 months: CMV Positive Donor: number analyzed (Participants) | 27 | 27
  36 months: CMV Positive Donor | 42 | 51
  36 months: CMV Negative Donor: number analyzed (Participants) | 15 | 14
  36 months: CMV Negative Donor | 20 | 28
  48 months: CMV Positive Donor: number analyzed (Participants) | 27 | 27
  48 months: CMV Positive Donor | 45 | 51
  48 months: CMV Negative Donor: number analyzed (Participants) | 15 | 14
  48 months: CMV Negative Donor | 21 | 28
  60 months: CMV Positive Donor: number analyzed (Participants) | 27 | 28
  60 months: CMV Positive Donor | 46 | 52
  60 months: CMV Negative Donor: number analyzed (Participants) | 15 | 15
  60 months: CMV Negative Donor | 21 | 29
  72 months: CMV Positive Donor: number analyzed (Participants) | 28 | 28
  72 months: CMV Positive Donor | 48 | 53
  72 months: CMV Negative Donor: number analyzed (Participants) | 15 | 15
  72 months: CMV Negative Donor | 21 | 29
  84 months: CMV Positive Donor: number analyzed (Participants) | 28 | 28
  84 months: CMV Positive Donor | 48 | 53
  84 months: CMV Negative Donor: number analyzed (Participants) | 15 | 15
  84 months: CMV Negative Donor | 21 | 31

42. Secondary Outcome: Creatinine Clearance at Month 24 and Every 12 Months up to Month 84
Description: Creatinine Clearance estimated by Cockcroft-Gault formula.
Time Frame: From Month 24 to Month 84
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Mean (Standard Deviation); unit: millimiters/minute
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Number analyzed (Participants) | 148 | 151
millimiters/minute
  24 months | 63.2 (23.85) | 62.9 (25.01)
  36 months | 63.9 (24.14) | 64.5 (25.33)
  48 months | 63.1 (23.81) | 62.6 (24.63)
  60 months | 62.2 (22.58) | 64.9 (27.85)
  72 months | 63.3 (28.98) | 64.7 (27.25)
  84 months | 59.5 (26.76) | 60.8 (25.39)

ADVERSE EVENTS:
Time Frame: Up to 7 years
Description: Analysis was performed on the safety analysis population. The safety population included all randomized participants.
Arm/Group | Valganciclovir CMV Prophylaxis | Pre-emptive CMV Therapy
Serious Adverse Events (participants affected / at risk) | 94/148 | 96/151
Other Adverse Events (participants affected / at risk) | 139/148 | 140/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir CMV Prophylaxis (N=148) | Pre-emptive CMV Therapy (N=151)
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 2 | 0
Lymphocele (Vascular disorders) | 6 | 4
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1
Prostatectomy (Surgical and medical procedures) | 1 | 0
Removal of ambulatory peritoneal catheter (Surgical and medical procedures) | 0 | 1
Ureteral stent removal (Surgical and medical procedures) | 0 | 1
Ureteric operation (Surgical and medical procedures) | 0 | 1
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kidney transplant rejection (Immune system disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 3
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 2
Acute psychosis (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 3 | 1
Graft complication (Injury, poisoning and procedural complications) | 0 | 2
Graft dysfunction (Injury, poisoning and procedural complications) | 0 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 2
Shunt blood flow excessive (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 3 | 0
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood calcium increased (Investigations) | 1 | 0
Blood creatinine abnormal (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 23 | 17
Blood glucose abnormal (Investigations) | 0 | 1
Blood parathyroid hormone increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 3 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Liver function test abnormal (Investigations) | 1 | 0
Occult blood positive (Investigations) | 0 | 1
Urine output decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Trifascicular block (Cardiac disorders) | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 5 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Benign intracranial hypertension (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Charles Bonnet syndrome (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Endophthalmitis (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Cupulolithiasis (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Sclerosing encapsulating peritonitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Postrenal failure (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0
Renal artery stenosis (Renal and urinary disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 3
Renal impairment (Renal and urinary disorders) | 3 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ureteral necrosis (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 2
Urinary fistula (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Abscess oral (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Endocarditis staphylococcal (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Gastroenteritis norovirus (Infections and infestations) | 1 | 1
Gastrointestinal infection (Infections and infestations) | 5 | 1
Graft infection (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 6
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 9 | 13
Urosepsis (Infections and infestations) | 1 | 7
Wound abscess (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir CMV Prophylaxis (N=148) | Pre-emptive CMV Therapy (N=151)
Hypertension (Vascular disorders) | 30 | 37
Hypotension (Vascular disorders) | 7 | 9
Fatigue (General disorders) | 5 | 11
Oedema (General disorders) | 27 | 31
Oedema peripheral (General disorders) | 34 | 30
Pain (General disorders) | 4 | 11
Pyrexia (General disorders) | 12 | 9
Insomnia (Psychiatric disorders) | 17 | 14
Sleep disorder (Psychiatric disorders) | 9 | 13
Blood creatinine increased (Investigations) | 23 | 21
Blood uric acid increased (Investigations) | 10 | 7
C-reactive protein increased (Investigations) | 13 | 11
Gamma-glutamyltransferase increased (Investigations) | 5 | 12
Anaemia (Blood and lymphatic system disorders) | 28 | 38
Hepatic enzyme increased (Investigations) | 14 | 7
Leukocytosis (Blood and lymphatic system disorders) | 7 | 9
Leukopenia (Blood and lymphatic system disorders) | 37 | 35
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Headache (Nervous system disorders) | 12 | 14
Tremor (Nervous system disorders) | 16 | 17
Abdominal pain upper (Gastrointestinal disorders) | 3 | 9
Constipation (Gastrointestinal disorders) | 13 | 15
Diarrhoea (Gastrointestinal disorders) | 41 | 42
Dyspepsia (Gastrointestinal disorders) | 5 | 8
Nausea (Gastrointestinal disorders) | 16 | 16
Vomiting (Gastrointestinal disorders) | 11 | 9
Haematuria (Renal and urinary disorders) | 8 | 8
Leukocyturia (Renal and urinary disorders) | 5 | 15
Proteinuria (Renal and urinary disorders) | 18 | 23
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 16
Acidosis (Metabolism and nutrition disorders) | 4 | 11
Diabetes mellitus (Metabolism and nutrition disorders) | 19 | 25
Glucose tolerance impaired (Metabolism and nutrition disorders) | 3 | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 17
Hypercholesterolaemia (Metabolism and nutrition disorders) | 17 | 16
Hyperkalaemia (Metabolism and nutrition disorders) | 15 | 20
Hyperlipidaemia (Metabolism and nutrition disorders) | 14 | 23
Hyperuricaemia (Metabolism and nutrition disorders) | 23 | 25
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 12 | 9
Metabolic acidosis (Metabolism and nutrition disorders) | 17 | 21
Bronchitis (Infections and infestations) | 6 | 8
Nasopharyngitis (Infections and infestations) | 36 | 34
Urinary tract infection (Infections and infestations) | 53 | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.